CLINICAL TRIAL: NCT00434018
Title: Enhancing Indoor, Community, and Advanced Wheelchair Skills in SCI
Brief Title: Enhancing Indoor, Community, and Advanced Wheelchair Skills in Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IIR 06-274
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Spinal Cord Injury
Keywords: Wheelchairs; Safety
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wheelchair Skills Training Program (Other): Subjects are provided with five weeks of wheelchair skills training, tailored to meet their needs. The WSP is a set of assessment and training protocols related to wheelchair skills. The WSP includes the Wheelchair Skills Test (WST), the Wheelchair Skills Training Program (WSTP) and related materials.
  Interventions: Behavioral: Wheelchair Skills Training
- Basic Health Education (Other): Basic health educational training sessions: Five sessions are held with subjects to provide them additional information regarding health related issues - such as nutrition, proper hand hygiene, sports, etc.
  Interventions: Behavioral: Basic Health Education

INTERVENTIONS:
Behavioral: Wheelchair Skills Training — Subjects are provided with five weeks of wheelchair skills training, tailored to meet their needs.
  Arms: Wheelchair Skills Training Program
Behavioral: Basic Health Education — Five sessions are held with subjects to provide them with educational information regarding health related issues - such as nutrition, proper hand hygiene, sports, etc.
  Arms: Basic Health Education

SUMMARY:
We propose to test an evidence-based wheelchair skills training program to optimize wheelchair safety and performance in veterans with SCI. The proposed training program incorporates emerging evidence on wheelchair biomechanics and motor-skills learning, and addresses recommendations in a new clinical practice guideline. Given the difficulty in translating wheelchair skills learned in a therapy clinic with "real world" problems in the home and community post-discharge, we are proposing to conduct the wheelchair skills training in and around the veteran's home. The immediate goal is to enhance ability, performance time, safety, community participation, and quality of life, while minimizing physical strain. The ultimate goal is to reduce morbidity/mortality associated with wheelchair use and promote successful aging with a disability.

DETAILED DESCRIPTION:
The purpose of this 3-year randomized controlled clinical trial is to evaluate use of a community-based wheelchair skills training program (WSTP). Objectives include:

1. Determine the immediate and sustained effects of a WSTP on ability, performance time, and physical strain.
2. Examine the effects of mediating and moderating variables on ability, performance time, and physical strain.
3. Examine the effects of a WSTP on safety, community participation, and quality of life.
4. Promote dissemination of WSTP in VA SCI Centers through two key activities: (a) Design innovative marketing plans to increase participation and promote patient-centeredness based on patient-perceived benefits. (b) Estimate health care resources needed to add home-based

ELIGIBILITY:
Inclusion Criteria:

* SCI for at least 1 year (neurologically stable)
* Level of injury: C6 and below who use manual wheelchair as a primary means of mobility
* Able to self-propel wheelchair
* Between the ages of 18-75
* Able to follow simple instructions

Exclusion Criteria:

* Progressive disease (e.g. spinal tumor)
* Extended bedrest for more than 30 days
* Ventilator-dependent
* Any cardiac or respiratory condition that would limit subject's physical performance
* Unstable medical conditions
* Use power wheelchair or scooter as primary means of mobility
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Groer, PhD MS, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (3):
- United States (3):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - VA Medical Center, Augusta, Augusta, Georgia
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment intervals at each site were as follows: 4/08-8/10 at Tampa, 6/08-8/10 at Boston, and 11/08-10/09 at Augusta. Recruitment efforts included posters in VA elevators and in clinic waiting rooms, study brochures, and/or referral of subject by primary care physicians.
Period: Overall Study
Arm/Group | Wheelchair Skills Training Program | Basic Health Education
Started | 69 | 69
Completed | 52 | 57
Not Completed | 17 | 12

BASELINE CHARACTERISTICS:
Population: One hundred thirty-eight veterans were recruited and randomly selected for group assignments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Wheelchair Skills Training Program | Basic Health Education | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.5) | 45.3 (13) | 45.7 (13.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 63 | 124
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 64 | 64 | 128
Region of Enrollment [Number; unit: participants]
  United States | 69 | 69 | 138

OUTCOME MEASURES:

1. Primary Outcome: Wheelchair Skills Test (WST)
Description: The WST is a standardized evaluation method that permits a set of representative wheelchair skills to be objectively, simply and inexpensively documented. The WST is an instrument for the objective evaluation of wheelchair skills. The WST consists of a series of commonly used wheelchair skills spanning the spectrum from those as basic as applying brakes to those as difficult as climbing curbs and performing wheelies. The WSC encompasses 57 skills (in Version 4.1) which result in a total score. The WST provide a pass-fail score for each skill. Refusal to attempt a skill (e.g. because of fear) constitutes a failing grade. The numerator is the Total Raw Score (i.e., the number of individual skills awarded a passing score) and the denominator is the number of applicable skills (i.e., the total number of skills minus those awarded NP scores). 100% is the maximum possible percentage score.
Time Frame: long term (1 year)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wheelchair Skills Training Program | Basic Health Education
Number analyzed (Participants) | 52 | 57
units on a scale | 90.4 (11.2) | 89.6 (11.7)
Statistical Analysis 1: Comparison: Wheelchair Skills Training Program vs Basic Health Education; Test type: Superiority or Other; p = 0.001, ANOVA

2. Secondary Outcome: Craig Handicap Assessment and Reporting Technique (CHART): Physical Independence Subscale
Description: Use as a measure of handicap that captures the interaction of the person and the environment, and of community reintegration and participation. The CHART quantifies handicap by evaluating five domains: physical independence, mobility, occupation, social integration, and economic self-sufficiency. The CHART is made up of 27 questions with responses that are countable or in a yes/no format. Each of the five subscales has a maximum score of 100, and they may be summed to form a total score. High scores indicate lesser handicap. The CHART was developed as a specific instrument to measure handicap, is the only measure of that concept validated specifically for persons with SCI, and is currently the most widely used measure related to community reintegration in SCI. The Physical Independence subscale measures the ability to sustain a customarily effective independent existence.
Time Frame: long term (1 year)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Basic Health Training: Basic health educational training sessions: Five sessions are held with subjects to provide them additional information regarding health related issues - such as nutrition, proper hand hygiene, sports, etc
Arm/Group | Wheelchair Skills Training Program | Basic Health Training
Number analyzed (Participants) | 52 | 57
units on a scale | 91 (19) | 91 (15)

3. Secondary Outcome: Craig Handicap Assessment and Reporting Technique (CHART): Mobility Subscale
Description: Use as a measure of handicap that captures the interaction of the person and the environment, and of community reintegration and participation. The CHART quantifies handicap by evaluating five domains: physical independence, mobility, occupation, social integration, and economic self-sufficiency. The CHART is made up of 27 questions with responses that are countable or in a yes/no format. Each of the five subscales has a maximum score of 100, and they may be summed to form a total score. High scores indicate lesser handicap. The CHART was developed as a specific instrument to measure handicap, is the only measure of that concept validated specifically for persons with SCI, and is currently the most widely used measure related to community reintegration in SCI. The Mobility Subscale measures the ability to move about effectively in his/her surroundings.
Time Frame: long term (1 year)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wheelchair Skills Training Program | Basic Health Training
Number analyzed (Participants) | 52 | 57
units on a scale | 93.7 (13.7) | 92.8 (11.4)

4. Secondary Outcome: Craig Handicap Assessment and Reporting Technique (CHART): Occupation Subscale
Description: Use as a measure of handicap that captures the interaction of the person and the environment, and of community reintegration and participation. The CHART quantifies handicap by evaluating five domains: physical independence, mobility, occupation, social integration, and economic self-sufficiency. The CHART is made up of 27 questions with responses that are countable or in a yes/no format. Each of the five subscales has a maximum score of 100, and they may be summed to form a total score. High scores indicate lesser handicap. The CHART was developed as a specific instrument to measure handicap, is the only measure of that concept validated specifically for persons with SCI, and is currently the most widely used measure related to community reintegration in SCI. The Occupation Subscale measures the ability to occupy time in the manner customary to that person's sex, age, and culture.
Time Frame: long term (1 year)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wheelchair Skills Training Program | Basic Health Training
Number analyzed (Participants) | 52 | 57
units on a scale | 75.1 (30.7) | 73.5 (29.8)

5. Secondary Outcome: Craig Handicap Assessment and Reporting Technique (CHART): Social Integration Subscale
Description: Use as a measure of handicap that captures the interaction of the person and the environment, and of community reintegration and participation. The CHART quantifies handicap by evaluating five domains: physical independence, mobility, occupation, social integration, and economic self-sufficiency. The CHART is made up of 27 questions with responses that are countable or in a yes/no format. Each of the five subscales has a maximum score of 100, and they may be summed to form a total score. High scores indicate lesser handicap. The CHART was developed as a specific instrument to measure handicap, is the only measure of that concept validated specifically for persons with SCI, and is currently the most widely used measure related to community reintegration in SCI. The Social Integration Subscale measures the ability to participate in and maintain customary social relationships.
Time Frame: long term (1 year)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wheelchair Skills Training Program | Basic Health Training
Number analyzed (Participants) | 52 | 57
units on a scale | 90 (15.7) | 90.5 (18.9)

6. Secondary Outcome: Craig Handicap Assessment and Reporting Technique (CHART): Economic Self-Sufficiency Subscale
Description: Use as a measure of handicap that captures the interaction of the person and the environment, and of community reintegration and participation. The CHART quantifies handicap by evaluating five domains: physical independence, mobility, occupation, social integration, and economic self-sufficiency. The CHART is made up of 27 questions with responses that are countable or in a yes/no format. Each of the five subscales has a maximum score of 100, and they may be summed to form a total score. High scores indicate lesser handicap. The CHART was developed as a specific instrument to measure handicap, is the only measure of that concept validated specifically for persons with SCI, and is currently the most widely used measure related to community reintegration in SCI. The Economic Self-Sufficiency subscale measures the ability to sustain customary socio-economic activity and independence.
Time Frame: long term (1 year)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wheelchair Skills Training Program | Basic Health Training
Number analyzed (Participants) | 52 | 57
units on a scale | 82.4 (33.9) | 86.5 (26.6)

ADVERSE EVENTS:
Time Frame: Study duration, up to 1 year.
Arm/Group | Wheelchair Skills Training | Basic Health Education
Serious Adverse Events (participants affected / at risk) | 8/69 | 5/69
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wheelchair Skills Training (N=69) | Basic Health Education (N=69)
Hospitalization due to infected ankle wound (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalization due to depression and acute alcohol Intoxication (General disorders) | 0 (0) | 1 (1)
Hospitalization due to chronic heel/knee ulcers and heavy alcohol consumption (General disorders) | 0 (0) | 1 (1)
Hospitalization due to fever and possible infection (General disorders) | 0 (0) | 1 (1)
Hospitalization due to pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization for colonoscopy screening (Investigations) | 1 (1) | 0 (0)
Hospitalization due to fever and nausea (General disorders) | 0 (0) | 1 (1)
Hospitalization due to fever and infection (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization due to bleeding colostomy and urinary tract infection (General disorders) | 0 (0) | 1 (1)
Hospitalization due to urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Hospitalization due to infected right foot pressure ulcer (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization due to bladder stone (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization due to wound re-opening (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization due to surgical incision re-opening (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization due to bladder biopsy and cystoscopy (Investigations) | 1 (1) | 0 (0)
Hospitalization due to emesis and dehydration (General disorders) | 1 (1) | 0 (0)
Hospitalization due to stroke/mental status change (General disorders) | 1 (1) | 0 (0)
Hospitalization due to fever and urinary tract infection (General disorders) | 1 (1) | 0 (0)
Hospitalization due to pneumonia and altered mental status (General disorders) | 1 (1) | 0 (0)
Hospitalization due to mental status change and dehydration (General disorders) | 1 (1) | 0 (0)
Hospitalized for fever and confusion (General disorders) | 1 (1) | 0 (0)
Hospitalized for pneumonia, leukocytosis, fever and UTI. (General disorders) | 1 (1) | 0 (0)
Hospitalized for mental status changes, vomiting blood and dehydration. (General disorders) | 1 (1) | 0 (0)
Hospitalized for fever, chills, and nephrostomy tube placement for kidney stone/IV anti (General disorders) | 1 (1) | 0 (0)
Hospitalization due to change in mental status and declining health (General disorders) | 1 (1) | 0 (0)
Hospitalization due to hand surgery. (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes